CLINICAL TRIAL: NCT04633473
Title: SIBTime: Media-enhanced Technology for Promoting the Behavioral Health and Family Relationships of Typically Developing Young Siblings
Brief Title: SIB-Time Web-application Tool for Typically Developing Siblings
Acronym: SIBTime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD015947
Record Dates: First submitted 2020-10-28; First posted 2020-11-18 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Family Relations; Sibling Relations
Keywords: Social Emotional Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIBTime (Experimental): 43 primary parents were assessed at enrollment, then provided the dual-language, media-enhanced SIBTime technology for 4 weeks, and then re-assessed at 4 weeks (after treatment completion).
  Interventions: Behavioral: SIB-Time Web-Application Tool

INTERVENTIONS:
Behavioral: SIB-Time Web-Application Tool — Parents used the dual-language SIBTime app to watch video stories about common sibling experiences, respond to question prompts, track connection routines, and listen to guided Acceptance and Commitment Therapy (ACT) exercises for parents. During the 4-week intervention period, parents used the app at their convenience.
  Other Names: SIBTime

SUMMARY:
In the United States, over 32.7 million people have special health, developmental, and mental health concerns. Most of these people have typically developing brothers and sisters. Across the lifespan, siblings share high levels of involvement in each other's lives, and also many of the concerns that parents of children with special needs experience, including isolation, a need for information, concerns about the future, and caregiving demands. Brothers and sisters also face issues that are uniquely theirs including emotions (resentment, worry, embarrassment, guilt), peer issues, and family communication challenges. The team of researchers, developers, and consultants built and tested an assistive media enhanced web-application tool for developing knowledge, skills, and routines for attending to TD siblings' (ages 3-5) social-emotional health and well-being.

DETAILED DESCRIPTION:
The investigators conducted a 4-week intervention to assess the English/Spanish, media-enhanced SIBTime web-application tool in terms of its relevance, acceptability, cultural appropriateness, and potential for efficacy to deliver a family-based intervention. The test used a within subjects pre-post design to detect changes in parent self-efficacy, family cohesion, and knowledge, and parent rating of sibling-parent relationship. Additionally, the investigators collected a post-test evaluation of consumer satisfaction and recommendations for modifications to the program.

ELIGIBILITY:
Inclusion Criteria

* Be the primary parent/guardian of a child with a disability
* Also be the primary parent/guardian of a typically developing child, 3-5 years old
* Speak English or Spanish
* Have access to a computer, tablet, or smartphone

Exclusion Criteria

• N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Vadasy, Ph.D., Principal Investigator — Oregon Research Behavioral Interventions Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were parents who were enrolled between 6/9/21 and 3/30/22. Participants were recruited through Advisory Board contacts, and social media.
Pre-assignment Details: Participants were parents who were enrolled in the study. Parents completed study measures. Parents engaged in activities with their child, but children were not enrolled and no data were collected from children.
Groups:
- SIBTime: 43 primary parents were assessed at enrollment, then provided the dual-language, media-enhanced SIBTime technology for 4 weeks, and then re-assessed at 4 weeks (after treatment completion).
  SIB-Time Web-Application Tool: Parents used the dual-language SIBTime app with their children. They watched video stories about common sibling experiences, responded to question prompts, tracked connection routines, and listened to guided ACT exercises for parents. During the 4-week intervention period, they used the app at their convenience.
Period: Overall Study
Arm/Group | SIBTime
Started | 43
Completed | 37
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- SIBTime: 43 primary parents were assessed at enrollment, then provided the dual-language, media-enhanced SIBTime technology for 4 weeks, and then re-assessed at 4 weeks (after treatment completion).
  SIB-Time Web-Application Tool: Parents used the dual-language SIBTime app with their children to watch video stories about common sibling experiences, respond to question prompts, track connection routines, and listen to guided ACT exercises for parents. During the 4-week intervention period, parents used the app at their convenience.
Arm/Group | SIBTime
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 43
Parent Demographic Form [Count of Participants; unit: Participants] | 43

OUTCOME MEASURES:

1. Primary Outcome: Parenting & Family Adjustment Scales (PAFAS) Parent/Child Relationship Subscale
Description: The Parenting & Family Adjustment Scales (PAFAS; Sanders et al., 2014) Parent/Child Relationship subscale measures the quality of the parent-child relationship, asking how true various statements have been over the past 4 weeks. The Parent/Child Relationship subscale is measured with 5 items, answered on a 5-point scale (0=Not at all; 4=Very much). Average scores range from 0 to 4, with higher scores indicating worse outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SIBTime: 43 primary parents were assessed at enrollment, then provided the dual-language, media-enhanced SIBTime technology for 4 weeks, and then re-assessed at 4 weeks (after treatment completion).
  SIB-Time Web-Application Tool: Parent-child dyads used the dual-language SIBTime app to watch video stories about common sibling experiences, respond to question prompts, track connection routines, and listen to guided Acceptance and Commitment Therapy (ACT) exercises for parents. During the 4-week intervention period, families used the app at their convenience.
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 0.26 (0.32)
  Posttest | 0.26 (0.35)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.922, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0

2. Primary Outcome: Parenting & Family Adjustment Scales (PAFAS) Parental Adjustment Subscale
Description: The Parenting & Family Adjustment Scales (PAFAS; Sanders et al., 2014) measures change in parenting practices, family cohesion, parent-child relationship quality, and parents' stress. The 30 items on the PAFAS sort into 7 subscales: Parental consistency, Coercive parenting, Positive encouragement, Parent-child relationship, Parental adjustment/stress, Family relationships, and Parental teamwork with partner. Items are rated on a 5-point scale (0-4) with higher scores worse.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 1.17 (0.71)
  Posttest | 1.07 (0.64)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.521, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.1

3. Primary Outcome: Parenting & Family Adjustment Scales (PAFAS) Family Relationships Subscale
Description: as for outcome 2
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 0.99 (0.59)
  Posttest | 0.94 (0.58)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.678, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.05

4. Primary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) Emotional Availability Subscale
Description: The Self-Efficacy for Parenting Tasks Index (SEPTI; Coleman & Karraker, 2000) - Emotional Availability subscale measures parents' self-efficacy for providing emotional support to their typically developing child and meeting their child's emotional needs. Parents rate their agreement or disagreement with a series of statements. The SEPTI Emotional Availability subscale is measured with 7 items. Respondents answer on a 6-point scale (1=Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SIBTime: 43 primary parents were assessed at enrollment, then provided the dual-language, media-enhanced SIBTime technology for 4 weeks, and then re-assessed at 4 weeks (after treatment completion).
  SIB-Time Web-Application Tool: Parent-child dyads used the dual-language SIBTime app to watch video stories about common sibling experiences, respond to question prompts, track connection routines, and listen to guided ACT exercises for parents. During the 4-week intervention period, families used the app at their convenience.
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 2.07 (0.69)
  Posttest | 1.93 (0.51)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.326, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.14

5. Primary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) Nurturance/Valuing/Empathic Responsiveness Subscale
Description: The Self-Efficacy for Parenting Tasks Index (SEPTI; Coleman & Karraker, 2000) - Nurturance/Valuing/Empathic Responsiveness subscale measures parents' self-efficacy for providing empathy, nurturance, and understanding to their typically developing child. Parents rate their agreement or disagreement with a series of statements. The SEPTI Nurturance/Valuing/Empathic Responsiveness subscale is measured with 8 items. Respondents answer on a 6-point scale (1=Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 1.93 (0.50)
  Posttest | 1.75 (0.37)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.09, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.18

6. Primary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) Play Subscale
Description: The Self-Efficacy for Parenting Tasks Index (SEPTI; Coleman & Karraker, 2000) - Play subscale measures parents' self-efficacy for playing with and having fun with their typically developing child. Parents rate their agreement or disagreement with a series of statements. The SEPTI Play subscale is measured with 7 items. Respondents answer on a 6-point scale (1=Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 2.98 (1.17)
  Posttest | 2.64 (0.89)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.154, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.34

7. Primary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) Teaching Subscale
Description: The Self-Efficacy for Parenting Tasks Index (SEPTI; Coleman & Karraker, 2000) - Teaching subscale measures parents' self-efficacy for explaining things and teaching their typically developing child about the world in a way that their child can understand. Parents rate their agreement or disagreement with a series of statements. The SEPTI Teaching subscale is measured with 9 items. Respondents answer on a 6-point scale (1=Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 2.39 (0.74)
  Posttest | 2.23 (0.68)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.309, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = -0.16

8. Primary Outcome: System Usability Scale (SUS)
Description: The System Usability Scale (SUS) is a commonly used 10-item measure (with a 5-point scale) of subjective perceptions of technology usability. To calculate the total SUS score, the responses to all 10 SUS questions are re-scaled and/or re-scored in a way that all items had values from zero to 4 with 4 being the most positive. These converted scores are added and then multiplied by 2.5 to convert the range of possible values 0-100 (instead of from 0 to 40). Higher scores are better.
Time Frame: Week 4
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 34
score on a scale | 81.99 (14.47)

9. Secondary Outcome: Engagement in Target Activities With Child - Frequency
Description: The Engagement in Target Activities with Child - Frequency subscale measures the frequency with which parents report engaging in specific "connection routine" activities with their typically developing child in the past month, across 17 items reflecting a range of program-targeted parenting behaviors. Respondents answer on a 7-point frequency scale (0=Never in the past month; 6=6 or more times per day); average scores range from 0 to 6, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 3.62 (0.80)
  Posttest | 3.88 (0.87)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.181, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0.26

10. Secondary Outcome: Engagement in Target Activities With Child - Self-efficacy
Description: The Engagement in Target Activities with Child - Self-Efficacy subscale measures parents' self-efficacy for engaging in specific "connection routine" activities with their typically developing child in the past month, across 17 items reflecting a range of program-targeted parenting behaviors. Respondents answer on a 10-point scale of how confident they are that they can carry out these behaviors (1=Not at all confident; 10=Highly confident); average scores range from 1 to 10, with higher scores indicating better outcomes.
Time Frame: Enrollment, and at 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SIBTime
Number analyzed (Participants) | 37
score on a scale
  Pretest | 7.65 (1.46)
  Posttest | 8.56 (1.10)
Statistical Analysis 1: Comparison: SIBTime; Test type: Superiority; p = 0.008, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0.91

11. Secondary Outcome: Family Usage of the SIBTime App - Number of Sessions
Description: Measure the families' usage of the SIBTime app using metrics and transcripts collected on the back-end database, including activation of the app; which elements are accessed; frequency, timing, and duration of engagements; and points of difficulty or failure.
Time Frame: At 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: Number of sessions
Arm/Group | SIBTime
Number analyzed (Participants) | 43
Number of sessions | 5.6 (4.2)

12. Secondary Outcome: Family Usage of the SIBTime App - Program Exposure
Description: as for outcome 11
Time Frame: At 4 weeks (after treatment completion)
Population: Primary parents of a child with a disability and a preschool age typically developing child.
Measure: Mean (Standard Deviation); unit: Percentage of program exposed to
Arm/Group | SIBTime
Number analyzed (Participants) | 43
Percentage of program exposed to | 69.9 (34.3)

ADVERSE EVENTS:
Time Frame: 1 month (4 weeks)
Description: All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not collected from parents.
Arm/Group | SIBTime
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT04633473/Prot_SAP_ICF_000.pdf